CLINICAL TRIAL: NCT05150743
Title: Using Longshi Scale and Barthel Index to Evaluate the Ability of Daily Living Activities in Stroke Survivors: a Comparative Study
Brief Title: Comparing the Responsiveness of Barthel Index and Longshi Scale in Assessing the ADL of Stroke Survivors
Status: Completed | Type: Observational
Sponsor: Shenzhen Second People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20210219006-FS01
Record Dates: First submitted 2021-10-09; First posted 2021-12-09 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2021-04

CONDITIONS: Disability Physical; Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The aim of this research was to compare the responsiveness of Barthel Index (BI) and Longshi Scale (LS) for assessing activities of daily living (ADL) in stroke survivors at different stage and we also aimed to observe changes of ADL score in stroke survivors over time.

DETAILED DESCRIPTION:
The whole experiment process has been supervised by a research assistant, and all the data collected are recorded on paper case report forms. The research assistant also takes charge of checking the consistency of data enter into the registry against predefined rules. Stroke survivors in Shenzhen Second People's Hospital have been invited to participate in this study and divide into three groups according to their duration of stroke (acute stroke, subacute stroke and chronic strike).

Data collection:

Baseline information was collected within 24 hours of admission. ADL of stroke survivors was assessed on admission, at discharge and 3 months after discharge.

Sample size calculation:

The sample size in this study was calculated according to the sample size calculation formula: n=[(µα+µβ)(µα+µβ)(1+1/k)p(1-p)]/(pe-pc)(pe-pc). Investigations in many places in China showed that varying degrees of dysfunction remain in 70%-80% of stroke survivors, and the disability rate is 30.2%-62.8%. In this reserach，p=(pe+kpc)/(1+k)，pe=0.3，pc =0.6, α=0.05，β=0.1, so µ0.05=1.6449，µ0.10=1.2816，thus the sample size in our study was n=47. We assume that 10% of them loss to follow-up, thus the sample size in our study was 52 in each group.

Statistical analysis:

1. Internal responsiveness First, standardized effect size (SES) was calculated by dividing the mean change in score between admission and discharge assessments by the standard deviation (SD) of the admission score. second, the standardized response mean (SRM) was obtained by dividing the mean change scores by the SD of the change score between admission and discharge scores. A value of SES or SRM>0.8 was large, 0.5 to 0.8 moderate, and 0.2 to 0.5 small.
2. External responsiveness The pearson correlation coefficient (r) was used to investigate the external responsiveness. An r value >0.75 represented good to excellent association; values of 0.50 to 0.75, moderate to good association; values of 0.25 to 0.50, fair association; and values ≤0.25, little association between the changes in scores on these measures. And the significance threshold was set at 0.05.
3. Receiver operating characteristic (ROC) curve For this study, the area under ROC curve (AUC) obtained by comparing subjects who improved by one or more levels on the modified Rankin scale vs. those who exhibit no change on the modified Rankin scale. Larger AUC means higher screening accuracy. In general, an AUC of 0.5 suggests no discrimination, 0.7 to 0.8 is considered acceptable, 0.8 to 0.9 is considered excellent, and more than 0.9 is considered outstanding.

ELIGIBILITY:
Inclusion Criteria:

* age 18-80 years
* diagnosis of cerebral infraction or intracerebral hemorrhage
* stable vital signs

Exclusion Criteria:

* brain tumor, Parkinson's disease or active epilepsy within three months
* impaired cognitive functions
* participation in any other clinical study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke survivors from the Department of Rehabilitation Medicine at Shenzhen Second People's Hospital are invited to participate in this study according to the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
The internal responsiveness of Longshi Scale at discharge | Baseline, 20 days after admission(discharge)
  The internal responsiveness of Longshi Scale is described using standardized effect size (SES) and the standardized response mean (SRM). Score of SES and SRM ranges from 0 to 1. Higher SES or SRM means better outcomes and SES or SRM > 0.5 is considered to be sufficient.
The internal responsiveness of Barthel Index at discharge | Baseline, 20 days after admission(discharge)
  The internal responsiveness of Barthel Index is described using SES and SRM. Score of SES and SRM ranges from 0 to 1. Higher SES or SRM means better outcomes and SES or SRM > 0.5 is considered to be sufficient.
The internal responsiveness of Longshi Scale at 3 months after discharge | Baseline, 3 months after discharge
  The internal responsiveness of Longshi Scale is described using standardized effect size (SES) and the standardized response mean (SRM). Score of SES and SRM ranges from 0 to 1. Higher SES or SRM means better outcomes and SES or SRM > 0.5 is considered to be sufficient.
The internal responsiveness of Barthel Index at 3 months after discharge | Baseline, 3 months after discharge
  The internal responsiveness of Barthel Index is described using SES and SRM. Score of SES and SRM ranges from 0 to 1. Higher SES or SRM means better outcomes and SES or SRM > 0.5 is considered to be sufficient.

SECONDARY OUTCOMES:
Pearson correlation coefficient (r) between Longshi Scale and Barthel Index at discharge | Baseline, 20 days after admission(discharge)
  The external responsiveness is described by Pearson correlation coefficient (r).
Pearson correlation coefficient (r) between Longshi Scale and Barthel Index at 3 months after discharge | Baseline, 3 months after discharge
  The external responsiveness is described by Pearson correlation coefficient (r).
Area under receiver operating characteristic curve of Longshi Scale at discharge | Baseline, 20 days after admission(discharge)
  The external responsiveness is described by area under receiver operating characteristic curve (AUC).
Area under receiver operating characteristic curve of Longshi Scale at 3 months after discharge | Baseline, 3 months after discharge
  The external responsiveness is described by area under receiver operating characteristic curve (AUC).
Area under receiver operating characteristic curve of Barthel Index at discharge | Baseline, 20 days after admission(discharge)
  The external responsiveness is described by area under receiver operating characteristic curve (AUC).
Area under receiver operating characteristic curve of Barthel Index at 3 months after discharge | Baseline, 3 months after discharge
  The external responsiveness is described by area under receiver operating characteristic curve (AUC).
Longshi Scale | Baseline, 20 days after admission(discharge) and 3 months after discharge
  A novel pictorial ADL assessment, 3-9 (better)
Barthel Index | Baseline, 20 days after admission(discharge) and 3 months after discharge
  ADL assessment, 0-100 (better)

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Second People's Hospital, Shenzhen, Gunagdong, China

IPD SHARING:
Plan to Share IPD: No
Contact the principal investigator for data if necessary